CLINICAL TRIAL: NCT03745274
Title: Randomised, Double-blind, Placebo-controlled, Phase I Dose- Escalation Study of Two Doses GHB04L1 in Healthy Adults
Brief Title: Two Doses of GHB04L1 for Pandemic Influenza Prophylaxis in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVIR Green Hills Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: GHB-CS02
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Influenza, Avian
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GHB04L1 (Experimental): GHB04L1 is administered as intranasal aerosol at a dose of 6.8 log10 or 7.5 log10 TCID50/dose/subject on day 1 and on day 29.
  Interventions: Biological: GHB04L1
- Placebo (Placebo Comparator): Placebo (buffer) is administered as intranasal aerosol on day 1 and on day 29.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GHB04L1 — Solution
  Arms: GHB04L1
Other: Placebo — Buffer solution
  Arms: Placebo

SUMMARY:
This study evaluates safety, tolerability and immunogenicity of two doses of GHB04L1, a liquid formulation of the replication- deficient influenza A/Vietnam/1203/04(H5N1)-like ∆NS1 virus in healthy adults. Subjects are randomised at a ratio of 2:1 for GHB04L1 (6.8 log10 or 7.5 log10 TCID50/dose/volunteer) or placebo.

DETAILED DESCRIPTION:
GHB04L1 is intended to provide a novel treatment approach for influenza virus H5N1 infection. Based on preclinical data from ferrets that demonstrated protection against challenge with wild-type virus following treatment with various dose levels of GHB04L1, vaccination with GHB04L1 might protect humans from influenza A (H5N1) virus infection.

Due to the lack of the NS1 protein, the ΔNS1 virus replicates efficiently in interferon-deficient cells but has lost its ability to grow in normal hosts and organisms. Immunisation with ΔNS1 mutant virus can cause only an abortive replication cycle in the nasal mucosa of vaccinated individuals. This allows development of replication-deficient intranasal vaccines with genetic stability of the attenuated phenotype and without virus shedding.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers, 18-50 years of age
* Seronegative for H5N1 (with antibody titres <1:10 detected in HAI assay)
* Seronegative for H1N1 (with antibody titres ≤1:20 detected in HAI assay)
* Written informed consent to participate in this study

Exclusion Criteria:

* Acute febrile illness (>37.0°C)
* Positive influenza immunoassay at baseline
* Signs of acute or chronic upper or lower respiratory tract illnesses (sneezing, cough, tonsillitis, otitis, etc.)
* History of severe atopy
* Influenza vaccination 2006/2007 and/or later
* Known increased tendency of nose bleeding
* Volunteers with clinically relevant abnormal paranasal anatomy
* Volunteers with clinically relevant abnormal laboratory values Females with positive urine pregnancy test prior to vaccination
* Simultaneous treatment with immunosuppressive drugs incl. corticosteroids (≥ 2 weeks) within 4 weeks prior to study medication application
* Clinically relevant history of renal, hepatic, GI, cardiovascular, haematological, skin, endocrine, neurological or immunological diseases
* History of leukaemia or cancer
* HIV or hepatitis B or C seropositivity
* Volunteers who had undergone rhino or sinus surgery or surgery of another traumatic injury of the nose within 30 days prior to application of study medication
* Volunteers who had received antiviral drugs, treatment with immunoglobulins or blood transfusions or an investigational drug within four weeks prior to study medication application
* Volunteers who had received anti-inflammatory drugs 2 days prior to study medication application
* Volunteers who were not likely to cope with the requirements of the study or with a significant physical or mental condition that may interfere with the completion of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12-19 (Actual); Primary Completion 2009-05-27 (Actual); Study Completion 2009-05-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | 8 weeks
  Occurrence of local and systemic adverse events overall and within 7 days after each study medication administration

SECONDARY OUTCOMES:
Viral shedding | 3 days
  Presence of GHB04L1 in mucosal samples from the nose
Local immune response | 8 weeks
  Local influenza A virus-specific immune response (IgA) in mucosal samples from the nose
Local cytokines response | 3 days
  Local cytokines response in mucosal samples from the nose
Systemic influenza A virus-specific antibody response | 8 weeks
  Systemic influenza A virus-specific antibody response determined by haemagglutination-inhibition assay (HAI) and micro-neutralisation assay (MNA) in serum samples
Systemic influenza A virus-specific T-cell response | 8 weeks
  Systemic influenza A virus-specific T-cell response determined by T-cell proliferation assay in blood samples
Systemic natural killer cell cytotoxicity | 5 weeks
  Systemic natural killer cell cytotoxicity in blood samples
Systemic T-cell Granzyme B assay | 8 weeks
  Systemic T-cell Granzyme B assay in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Kiselev, Prof, Principal Investigator — Research Institute of Influenza, Russian Academy of Medical Sciences
Locations (1):
- Research Institute of Influenza, Russian Academy of Medical Sciences, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicolodi C, Groiss F, Kiselev O, Wolschek M, Seipelt J, Muster T. Safety and immunogenicity of a replication-deficient H5N1 influenza virus vaccine lacking NS1. Vaccine. 2019 Jun 19;37(28):3722-3729. doi: 10.1016/j.vaccine.2019.05.013. Epub 2019 May 30. PMID 31155415